CLINICAL TRIAL: NCT04540575
Title: Reducing Disparity in Receipt of Mother's Own Milk in Very Low Birth Weight Infants: An Economic Intervention to Improve Adherence to Sustained Maternal Breast Pump Use
Brief Title: Reducing Disparity in Receipt of Mother's Own Milk in Very Low Birth Weight Infants
Acronym: ReDiMOM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 18060410; R01MD013969 (NIH)
Record Dates: First submitted 2020-08-19; First posted 2020-09-07 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Pumping, Breast; Milk, Human; Infant, Very Low Birth Weight; Preterm Birth
Keywords: Race/ethnicity; Mother's Own Milk; Disparity; Economic
MeSH Terms: conditions — Breast Milk Expression; Premature Birth

STUDY DESIGN:
Intervention Model Description: Mothers will be randomized into one of two groups after enrollment. Group 1, or "Mother Provides Mother's Own Milk (MOM)", will receive the standard of care. Group 2, or "NICU Acquires MOM", will receive the intervention. Two levels based on gestational age (extremely preterm < 28 weeks vs. very preterm 28-31 6/7 weeks, with approximately 50% expected in each group based on historical Rush University NICU births) will be crossed with three racial/ethnic categories (black, Hispanic, and white). The stratified random allocation table will be integrated into the baseline demographic questionnaire programmed in REDCap, allowing both patient and interviewer to be blind to condition until the end of the consent process and interview.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mother Provides MOM (Active Comparator): Receive Rush NICU standard of care lactation support
  Interventions: Behavioral: Mother Provides MOM
- NICU Acquires MOM (Experimental): Receive economic interventions in addition to Rush NICU standard of care lactation support
  Interventions: Behavioral: NICU Acquires MOM; Behavioral: Mother Provides MOM

INTERVENTIONS:
Behavioral: NICU Acquires MOM — Mother receives 1) hospital-grade electric smart breast pump for home use at no charge to the mother while the infant is in the NICU and the mother continues to pump; 2) free pickup of expressed MOM from home to transport to NICU 2-3 times per week during weekdays as needed; 3) receives payment for opportunity costs of pumping and handling milk at $24.00/day for each day that the mother pumps during her infant's NICU stay
  Arms: NICU Acquires MOM
Behavioral: Mother Provides MOM — Mother receives standard Rush NICU lactation care

SUMMARY:
In the US, the burden of very low birth weight (VLBW; <1500 g) birth is borne disproportionately by black (non-Hispanic black/African American) mothers who are 2.2-2.6 times more likely than nonblack mothers to deliver VLBW infants. This disparity is amplified because black VLBW infants are significantly less likely to receive mother's own milk (MOM) feedings from birth until neonatal intensive care unit (NICU) discharge than nonblack infants, which adds to the lifelong burden of VLBW birth with increased risk of morbidities and greater costs. Pumping is associated with out-of-pocket and opportunity costs that are borne by mothers, unlike donor human milk and formula, which are paid for by NICUs.

This innovative trial will determine the effectiveness of the intervention in reducing the disparity in MOM feedings and provide an economic analysis of the interventions, yielding critical data impacting generalizability and likelihood of implementation of results. The investigators hypothesize that mothers who receive intervention will have greater pumping volume and duration and their infants will be more likely to receive MOM at NICU discharge compared to mothers who receive standard of care lactation care and their infants.

DETAILED DESCRIPTION:
In the US, the burden of very low birth weight (VLBW; <1500 g) birth is borne disproportionately by black (non-Hispanic black/African American) mothers who are 2.2-2.6 times more likely than nonblack mothers to deliver VLBW infants. This disparity is amplified because black VLBW infants are significantly less likely to receive mother's own milk (MOM) feedings from birth until neonatal intensive care unit (NICU) discharge than nonblack infants, which adds to the lifelong burden of VLBW birth with increased risk of morbidities and greater costs. Even though black mothers of VLBW infants initiate MOM provision at rates similar to nonblack mothers and have similar goals to sustain MOM provision through to NICU discharge, there is a significant disparity in MOM feedings at NICU discharge. Only the mother can mitigate the disparity in MOM feedings at NICU discharge for the VLBW infant by: 1) sustaining breast pump use (6-8 times/day) for the entire NICU hospitalization (average = 73 days), and 2) transporting the MOM that is pumped in the home to the NICU for infant feedings. Pumping is associated with out-of-pocket and opportunity costs that are borne by mothers, unlike donor human milk and formula, which are paid for by NICUs.

The ReDiMOM randomized controlled trial will implement and evaluate an intervention (NICU acquires MOM) developed to offset the aforementioned costs that serve as barriers to sustaining MOM feedings. The intervention includes free hospital-grade electric breast pump, pickup of MOM, and payment for opportunity costs. The intervention will be evaluated in comparison to the current standard of care (mother provides MOM). Data will be collected from several sources including REDCap surveys, data extraction from the electronic medical record and hospital decision support/financial cost accounting system, smart breast pump data and measurement of pumped MOM volume.

This innovative trial will determine the effectiveness of the intervention in reducing the disparity in MOM feedings and provide an economic analysis of the interventions, yielding critical data impacting generalizability and likelihood of implementation of results. The investigators hypothesize that mothers who receive intervention will have greater pumping volume and duration and their infants will be more likely to receive MOM at NICU discharge compared to mothers who receive standard of care lactation care and their infants.

ELIGIBILITY:
Inclusion Criteria:

* MATERNAL: Delivery, or anticipated delivery, of infant with gestational age < 32 0/7 weeks at Rush, age ≥18 years, US citizen or legal resident, fluent in English or Spanish
* INFANT: Birth gestational age (GA)< 32 0/7 weeks, no significant congenital anomalies or chromosomal defects, <144 hours of age at enrollment, multiples may be included

Exclusion Criteria:

* Mothers with health conditions that are incompatible with milk provision per the clinical judgment of the NICU attending caring for the infant, mother is less than 18 years of age, mother has participated in this study with a previous pregnancy, mother is enrolled in another study that impacts lactation, in the neonatologist's opinion the infant is unlikely to survive, or mother is coronavirus (COVID-19) positive and unable to visit the NICU due to quarantine or infection-control requirements during the 144-hour post-delivery randomization window.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 611 (Estimated)
Dates: Start 2020-12-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Receipt of MOM at NICU Discharge | Through study completion, an average of 10 weeks
  Determined from the last full day of hospitalization and categorized as "Yes" if the infant received any or exclusive MOM and "No" if the infant received only formula.

SECONDARY OUTCOMES:
Receipt of any MOM | Through study completion, an average of 10 weeks
  Determined from the entire hospitalization and categorized as "Yes" if the infant received any or exclusive MOM and "No" if the never received MOM during the hospitalization.
Duration of MOM feedings | Through study completion, an average of 10 weeks
  Determined from the entire hospitalization and calculated as the number of days infant received any MOM.
Cumulative dose of MOM feedings | Through study completion, an average of 10 weeks
  Determined from the entire hospitalization and calculated as the total volume of MOM received by the infant.
Duration of MOM pumped | Through study completion, an average of 10 weeks
  Determined from the entire hospitalization and calculated as the number of days mother pumped MOM.
Volume of MOM pumped | Through study completion, an average of 10 weeks
  Determined from the entire hospitalization and calculated as the total volume of MOM pumped by the mother.
Healthcare system costs | Through study completion, an average of 10 weeks
  Costs borne by healthcare providers or third-party payers, including the cost of the hospital stay and donor human milk and formula costs.
Participant costs in US Dollars | Through study completion, an average of 10 weeks
  Participant costs will be measured in dollars and will be the sum of opportunity costs (i.e., mother's time spent pumping (mothers in control group only), time off work to visit NICU), caregiving costs for other children or adults when mother or partner visits the NICU, transportation costs, lodging costs, and other out-of-pocket costs
ReDiMOM Intervention Costs in US Dollars | Through study completion, an average of 10 weeks
  The costs of the intervention including milk pick-up, free provision of pumps, and opportunity costs payments for the intervention arm.

CONTACTS AND LOCATIONS:
Overall Officials: Aloka L Patel, MD, Principal Investigator — Rush University Medical Center, Department of Pediatrics; Tricia J Johnson, PhD, Principal Investigator — Rush University Medical Center, Department of Health Systems Management
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification
Supporting Information: Study Protocol, ICF
Time Frame: 2 to 5 years after publication of final results
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose and scientifically appropriate per the ReDiMOM principal investigators.

REFERENCES:
- [Background] Johnson TJ, Patel AL, Bigger HR, Engstrom JL, Meier PP. Economic benefits and costs of human milk feedings: a strategy to reduce the risk of prematurity-related morbidities in very-low-birth-weight infants. Adv Nutr. 2014 Mar 1;5(2):207-12. doi: 10.3945/an.113.004788. PMID 24618763
- [Background] Patel AL, Schoeny ME, Hoban R, Johnson TJ, Bigger H, Engstrom JL, Fleurant E, Riley B, Meier PP. Mediators of racial and ethnic disparity in mother's own milk feeding in very low birth weight infants. Pediatr Res. 2019 Apr;85(5):662-670. doi: 10.1038/s41390-019-0290-2. Epub 2019 Jan 18. PMID 30679795
- [Background] Patra K, Hamilton M, Johnson TJ, Greene M, Dabrowski E, Meier PP, Patel AL. NICU Human Milk Dose and 20-Month Neurodevelopmental Outcome in Very Low Birth Weight Infants. Neonatology. 2017;112(4):330-336. doi: 10.1159/000475834. Epub 2017 Aug 3. PMID 28768286
- [Background] Jegier BJ, Johnson TJ, Engstrom JL, Patel AL, Loera F, Meier P. The institutional cost of acquiring 100 mL of human milk for very low birth weight infants in the neonatal intensive care unit. J Hum Lact. 2013 Aug;29(3):390-9. doi: 10.1177/0890334413491629. Epub 2013 Jun 17. PMID 23776080
- [Background] Profit J, Gould JB, Bennett M, Goldstein BA, Draper D, Phibbs CS, Lee HC. Racial/Ethnic Disparity in NICU Quality of Care Delivery. Pediatrics. 2017 Sep;140(3):e20170918. doi: 10.1542/peds.2017-0918. PMID 28847984
- [Background] Trang S, Zupancic JAF, Unger S, Kiss A, Bando N, Wong S, Gibbins S, O'Connor DL; GTA DoMINO Feeding Group. Cost-Effectiveness of Supplemental Donor Milk Versus Formula for Very Low Birth Weight Infants. Pediatrics. 2018 Mar;141(3):e20170737. doi: 10.1542/peds.2017-0737. PMID 29490909
- [Background] Krubiner CB, Merritt MW. Which strings attached: ethical considerations for selecting appropriate conditionalities in conditional cash transfer programmes. J Med Ethics. 2017 Mar;43(3):167-176. doi: 10.1136/medethics-2016-103386. Epub 2016 Oct 5. PMID 27707877
- [Background] Belfort MB, Anderson PJ, Nowak VA, Lee KJ, Molesworth C, Thompson DK, Doyle LW, Inder TE. Breast Milk Feeding, Brain Development, and Neurocognitive Outcomes: A 7-Year Longitudinal Study in Infants Born at Less Than 30 Weeks' Gestation. J Pediatr. 2016 Oct;177:133-139.e1. doi: 10.1016/j.jpeds.2016.06.045. Epub 2016 Jul 29. PMID 27480198
- [Background] Relton C, Strong M, Thomas KJ, Whelan B, Walters SJ, Burrows J, Scott E, Viksveen P, Johnson M, Baston H, Fox-Rushby J, Anokye N, Umney D, Renfrew MJ. Effect of Financial Incentives on Breastfeeding: A Cluster Randomized Clinical Trial. JAMA Pediatr. 2018 Feb 5;172(2):e174523. doi: 10.1001/jamapediatrics.2017.4523. Epub 2018 Feb 5. PMID 29228160
- [Background] Washio Y, Humphreys M, Colchado E, Sierra-Ortiz M, Zhang Z, Collins BN, Kilby LM, Chapman DJ, Higgins ST, Kirby KC. Incentive-based Intervention to Maintain Breastfeeding Among Low-income Puerto Rican Mothers. Pediatrics. 2017 Mar;139(3):e20163119. doi: 10.1542/peds.2016-3119. Epub 2017 Feb 6. PMID 28167511
- [Derived] Johnson TJ, Meier PP, Schoeny ME, Bucek A, Janes JE, Kwiek JJ, Zupancic JAF, Keim SA, Patel AL. Study protocol for reducing disparity in receipt of mother's own milk in very low birth weight infants (ReDiMOM): a randomized trial to improve adherence to sustained maternal breast pump use. BMC Pediatr. 2022 Jan 7;22(1):27. doi: 10.1186/s12887-021-03088-y. PMID 34996401